CLINICAL TRIAL: NCT01202318
Title: Pilot Prospective Cohort to Determine the Comparative Diagnostic Accuracy of Card 28 to Card 28 and Cincinnati Stroke Scale.
Brief Title: Comparative Evaluation of Stroke Triage Algorithms for Emergency Medical Dispatchers
Acronym: MeDS
Status: Withdrawn | Type: Observational
Why Stopped: The study design was changed to a prospective cohort study due to difficulties in using a randomized approach in an emergency setting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H60373-35400-01
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
Keywords: Cerebrovascular Accident; Stroke,Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will compare the diagnostic accuracy of Card 28 stroke protocol to Card 28 and Cincinnati Stroke Scale, when used by emergency medical dispatchers to interrogate a 911 call suggestive of stroke.

The authors hypothesize that a combination of Card 28 plus the Cincinnati Stroke Scale (CSS) will improve the diagnostic accuracy of emergency medical dispatchers for stroke.

ELIGIBILITY:
Inclusion Criteria:

1. All 911 calls transferred by local Public Service Answering Points (PSAPs) to the County Communication center of Santa Clara County where the emergency medical dispatchers complete the interrogation using MPDS protocols.
2. All 911 calls received directly at the County Communication center of Santa Clara County where emergency medical dispatchers complete the interrogation using the MPDS protocols.
3. All 911 calls received from subjects (patient) aged > 18 years or second party calls (by-stander or family who are in close proximity to the patient and can administer the tool) by subjects > 18 years of age.

Exclusion Criteria:

1. All calls that require immediate response (ECHO level determinant for life threatening conditions) and emergency medical dispatchers cannot complete Card 28
2. Calls answered by emergency medical dispatchers who have not completed training on the use of Cincinnati Stroke Scale.
3. Calls originating from the cities of Palo Alto, Mountain View, Sunnyvale, Santa Clara, and San Jose that are not interrogated by the County Communication Center for Santa Clara County.
4. 911 calls with no available outcomes in the final discharge database.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population consists of all 911 callers with symptoms suggestive of stroke in the participating county. Specifically, the accessible population for this study is the group of patients whose 911 calls are answered and interrogated by the emergency medical dispatchers at the County Communication Center, Santa Clara.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prasanthi Govindarajan, MBBS, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- Alameda County, Alameda, California, United States